CLINICAL TRIAL: NCT01111864
Title: The Effect of Iron Fortification of Complementary Foods on Iron Status and Infant Gut Microbiota in Kenya
Brief Title: Changes in Microbiota and Iron Status After Iron Fortification of Complementary Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of KwaZulu (Other); University of Nairobi (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2-cercamondi
Record Dates: First submitted 2010-04-23; First posted 2010-04-28 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Iron; Micronutrients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MixMe powder (iron & micronutrients) (Experimental)
  Interventions: Dietary Supplement: fortification with iron and micronutrients
- MixMe powder (micronutrients, no iron) (Placebo Comparator)
  Interventions: Dietary Supplement: fortification with iron and micronutrients
- Sprinkles (iron and micronutrients) (Experimental): Vitamin A 300 µg; Vitamin C 30 mg; Folic Acid 160 µg; Iron 12.5 mg; Zinc 5 mg
  Interventions: Dietary Supplement: Sprinkles
- Sprinkles (micronutrients, no iron) (Placebo Comparator): Vitamin A 300 µg; Vitamin C 30 mg; Folic Acid 160 µg; Zinc 5 mg
  Interventions: Dietary Supplement: Sprinkles

INTERVENTIONS:
Dietary Supplement: fortification with iron and micronutrients — Iron 0 or 2.5 mg; Copper 0.34 mg; 30 µg Iodine; 7 µg Selenium; 2.5 mg Zinc; 100 µg Vitamin A; Vitamin D 5 µg; 5 mg Tocopherol Equivalent; 30 µg Vitamin K1; 10.5 mg Thiamine; 0.5 mg Riboflavin; 0.5 mg Pyridoxine; 90 µg Folic Acid Anhydrous; 6 mg Niacinamide; 60 mg Vitamin C; 0.9 µg Vitamin B12
  Arms: MixMe powder (iron & micronutrients); MixMe powder (micronutrients, no iron)
Dietary Supplement: Sprinkles — Daily 12.5mg Ferrous fumarate iron with microntrient is compared to no iron with micronutrients. Duration of intervention is 4 months, 80 infants will be inclulded.
  Arms: Sprinkles (iron and micronutrients); Sprinkles (micronutrients, no iron)

SUMMARY:
Infants and children under two years are the group with the highest rates of iron deficiency anemia. Provision of sufficient dietary iron to this age group is a challenge, and in-home iron fortification of complementary foods using micronutrient powders can be an effective approach. However, WHO has recently cautioned against untargeted use of in-home micronutrient powders that contain the entire iron RDA for a child in a single dose in areas with high rates of infections from malaria and diarrheal disease. Therefore, in this study, we will investigate the effect on the infant gut microbiota of a low dose (ca. 25% of the RDA) of highly bioavailable iron, provided by a micronutrient powder added to a complementary food.

The study aim is to determine if in-home fortification using an iron-containing micronutrient powder in Kenyan infants will improve iron status and/or modify the composition and metabolic activity of the gut microbiota. Active surveillance will be done weekly to monitor the health of the infants.

Our study will be done in a subgroup (n=160) of a larger double-blind controlled feeding trial in which 330 infants will be randomized to receive a micronutrient powder containing either 2.5 mg iron or no iron for 1 year. In our substudy, the infants will be studied only over the first 6 months of the 1 year intervention. Blood samples, taken at baseline and after 6 months will be used to define the iron status and the anemia level of the infants. Stool samples (2 at baseline before intervention, 6 throughout the study and additional samples in case of diarrhea) will be obtained for analysis of the gut microbiota. In the entire study (n=330), we will measure changes in iron status over 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Mother at least ≥15 years of age, infants 5.5- 6.5 months
* Willingness to provide informed consent
* Apparent good health
* Long-term residence in study site and anticipating residing in the area for at least 3 years
* Speak a Mjikenda language or Kiswahili in the home
* Willingness to provide blood samples during clinic visits

Exclusion Criteria:

* Hemoglobin <70 g/L for infants; these infants will be referred for treatment at the local health clinic/hospital.
* Acute or chronic pulmonary, cardiovascular, hepatic, renal or neurological condition or any other finding that in the opinion of the PI or co-researchers that would increase risk of participating in the study.
* Other conditions that in the opinion of the PI or co-researchers would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol

Ages: 24 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2010-02; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
gut microbiota composition | Fecal sample after 2 months
  Changes in gut microbiota composition

SECONDARY OUTCOMES:
iron status | 12 months
  Efficacy of iron fortification in complementary foods

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, M.D., Study Director — Human Nutrition Laboratory, Swiss Federal Institute of Technology; Jane Kvalsvig, PhD, Principal Investigator — Department of Public Health Medicine, Nelson Mandela School of Medicine, South Africa
Locations (1):
- Kikoneni Clinic, Kikoneni, Kwale County, Kenya

REFERENCES:
- [Derived] Jaeggi T, Kortman GA, Moretti D, Chassard C, Holding P, Dostal A, Boekhorst J, Timmerman HM, Swinkels DW, Tjalsma H, Njenga J, Mwangi A, Kvalsvig J, Lacroix C, Zimmermann MB. Iron fortification adversely affects the gut microbiome, increases pathogen abundance and induces intestinal inflammation in Kenyan infants. Gut. 2015 May;64(5):731-42. doi: 10.1136/gutjnl-2014-307720. Epub 2014 Aug 20. PMID 25143342